CLINICAL TRIAL: NCT02306837
Title: A Phase II Trial of Consolidation Chemothetapy for Patients With Relapse or Refractory Lymphoid Malignancies After Autologous Stem Cell Transplantation
Brief Title: Consolidation Chemotherapy After Autologous Stem Cell Transplantation for Lymphoid Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation Center, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lym-Auto-RJH-2014
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Effects of Chemotherapy
Keywords: lymphoma, consolidation chemotherapy, auto-HSCT
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Consolidation chemo (Experimental): Patients recieved 3 cycles of consolidation chemotherapy post-auto-HSCT: mini-Bu-Cy-E regimen
  Interventions: Drug: Bu-CY-E

INTERVENTIONS:
Drug: Bu-CY-E — mini Bu-Cy-E as consolidation chemotherapy after autologous HSCT
  Other Names: mini Bu-Cy-E

SUMMARY:
To imporve the outcome of patients with relapsed/refractory lymphoma, we conduct a clinical trial to test the efficacy and feasibility of consolidation chemotherapy after autologous stem cell transplantation

DETAILED DESCRIPTION:
Patients with relapsed or refractory lymphoma will be included. All patients will undergo PBSC mobilization with CTX and G-CSF. After sucessful collection of CD34+ over 1x109/L, autologous stem cel ltransplantation with Bu-Cy-E conditioning will be given. Two months after auto-HSCT, a PET-CT will be performed and all patients with CR, CRu and PR will recieved 3 cycles of mini-Bu-Cy-E as consolidation 3, 6 and 9 months after auto-HSCT. For patients with SD or PD after auto-HSCT will refered to the allogeneic transplantatio program and take off the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refracotry NHL or HD: PR or SD after first line salvage chemotherapy;
* ECOG: 0-2
* Tbil < 1.5x ULN and AST/ALT <2.5x ULN
* With informed consent

Exclusion Criteria:

* Life expectancy < 3 months
* Women in pregnancy
* uncontrollable infection disease
* serum Cr >400mmol/l
* uncontroled diabetis and heart disease

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2-year

SECONDARY OUTCOMES:
overall survival | 2-year
progression | 2-year
  PET-CT measurement
transplantation-related mortality | 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Hu, M.D,, Principal Investigator — Rui Jin Hospital, Shanghai Jiaotong Unic\versity School of Medicine
Locations (2):
- China (2):
  - Rui Jin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai
  - Shanghai No 10 Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided